CLINICAL TRIAL: NCT02978053
Title: The Effects of Bright Light on Adaptation to Night Work Among Nurses
Brief Title: Light Treatment to Shift-working Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Bjorn Bjorvatn, Professor, University of Bergen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UiB112016
Record Dates: First submitted 2016-11-25; First posted 2016-11-30 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Shift-Work Sleep Disorder
Keywords: Bright light; Sleepiness; Sleep; Psychomotor vigilance
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleepiness | interventions — Red Light

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright light (Experimental): 10 000 lux
  Interventions: Behavioral: Bright light
- Red light (Placebo Comparator): 400 lux
  Interventions: Behavioral: Red light

INTERVENTIONS:
Behavioral: Bright light — Bright light for 30 minutes during night shifts (between 2 AM and 3 AM the first night, between 3 AM and 4 AM the second night, between 4 AM and 5 AM the third night).
  Arms: Bright light
Behavioral: Red light — Red light for 30 minutes during night shifts (between 2 AM and 3 AM the first night, between 3 AM and 4 AM the second night, between 4 AM and 5 AM the third night).
  Arms: Red light

SUMMARY:
This project examines 1) the effects of appropriately timed bright light on adaptation (in terms of sleep and sleepiness) to three consecutive night shifts; and 2) the effects of such bright light on re-adaptation (in terms of sleep and sleepiness) to a day-oriented schedule after the night shift period.

DETAILED DESCRIPTION:
Shift workers frequently experience sleepiness during night shifts, which may have consequences for performance. Sleep duration is often shortened after a night shift. Properly timed bright light treatment is efficient in delaying the circadian rhythm and can enhance alertness, increase performance and prolong sleep after night shifts. There is a lack of studies on light treatment to rotating shift workers. This study is a randomized controlled crossover trial evaluating the effect of bright light treatment on sleep and sleepiness in rotating shift workers with three consecutive night shifts. The aim is to evaluate whether bright light treatment improves adaptation to three consecutive night shifts (reduces sleepiness during night shifts and improves sleep after night shifts), as well as whether such treatment affects re-adaptation to a day-oriented schedule after the night shift period.

ELIGIBILITY:
Inclusion Criteria:

* A rotating shift work schedule involving three days without night shifts, followed by three consecutive night shifts, followed by three days without night shifts
* Problems with sleepiness during night shifts

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Sleepiness during the night shifts | 3 days
  Self-reported using the Karolinska Sleepiness Scale (KSS)

SECONDARY OUTCOMES:
Psychomotor vigilance during night shifts | 3 days
  Objective data from a 5 min computer based psychomotor vigilance test (PC-PVT) taken once during each night shift
Sleep after the night shifts | 3 days
  Self-reported using a sleep diary; objective data from actigraphs
Sleepiness during the days after the night shift period | 3 days
  Self-reported using the Karolinska Sleepiness Scale (KSS)
Sleep during the days after the night shift period | 3 days
  Self-reported using a sleep diary; objective data from actigraphs
Functioning on each shift, and shift period in total, compared to under normal conditions | 6 days
  Self-reported perception of effect of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Bjorvatn, MD, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No